CLINICAL TRIAL: NCT05595447
Title: Rescue With Brentuximab Plus PD-1 Blockade Followed by Autotransplantation and Consolidation With Brentuximab Plus PD-1 Blockade in Patients With Relapsed/Refractory Hodgkin Lymphoma: Exploratory Single-arm Analysis
Brief Title: Treatment Strategy for Relapsed/Refractory Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Regional de Alta Especialidad del Bajio (Other)
Collaborators: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Lauro Fabian Amador Medina, Principal Investigator, Hospital Regional de Alta Especialidad del Bajio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI/HRAEB/038/2022
Record Dates: First submitted 2022-10-19; First posted 2022-10-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-12

CONDITIONS: Hodgkin Lymphoma; Refractory Hodgkin Lymphoma; Relapsed Hodgkin's Disease, Adult
Keywords: refractory; relapsed; hodgkin lymphoma
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — Brentuximab Vedotin; Nivolumab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Brentuximab plus PD-1 blocked x 8 plus ASCT (PEAM condicioning) plus maintanance Brentuximab plus PD-1 x 8 cycles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brentuximab plus PD-1 blocked plus ASCT plus maintenance Brentuximab plus PD-1 (Experimental): Brentuximab plus PD-1 blocked x 8 cycles plus ASCT plus maintenance Brentuximab plus PD-1 x 8 cycles
  Interventions: Drug: Brentuximab Vedotin 50 MG [Adcetris]

INTERVENTIONS:
Drug: Brentuximab Vedotin 50 MG [Adcetris] — Brentuximab plus blocked PD-1 plus ASCT plus maintenance Brentuximab plus blocked PD-1
  Other Names: Nivolumab; Pembrolizumab

SUMMARY:
The choice of the best second-line therapy in patients with high LH R/R risk, it is a niche of knowledge not covered at the moment, especially the role of Brentuximab (BV) plus PD-1 blockade and auto-HSCT.

What is the progression-free survival and rate of metabolic responses complete in patients with high-risk R/R HL with the treatment strategy: BV+ PD-1 blockade consolidation with Auto-HSCT and maintenance with BV + PD-blockade

1?

DETAILED DESCRIPTION:
Patientes with Refractory/relapsed Hodgkin Lymphoma (HL R/R) with multiple failed therapies represent a therapeutic dilemma. The goal of next-line treatment is long-term disease control with manageable adverse reactions. Given the limited therapeutic options for patients with HL R/R, better therapies should be sought, more effective, with better tolerability, less toxicity, with increased overall survival (OS) of the patients, with the aim of improving outcomes in terms of disease-free survival progression (PFS) of the current standard treatment. Since currently only 50% of the patients with high-risk R/R HL treated with the standard regimen achieve healing. The high effectiveness and low toxicity of immunotherapy with prolonged remission or stabilization of the disease make it a new treatment option promising for HL R/R. Based on the above, a treatment strategy is proposed to rescue base with Brentuximab plus PD-1 blockade followed by autotransplantation and consolidation with Brentuximab plus PD-1 blockade in patients with Hodgkin lymphoma High-Risk Relapse/Refractory Compared to Reported OS and PFS Rates in the literature obtained with standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed/refractory Hodgkin lymphoma to ABVD with definition of high risk.
2. Age ≥ 18 years and ≤ 90 years.
3. Adequate liver function, defined as:

   * Total serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * Serum aspartate aminotransferase (AST) ≤ 3.0 x ULN
   * Serum alanine aminotransferase (ALT) ≤ 3.0 x ULN
4. Adequate renal functions, defined as:

   • Serum creatinine ≤ 1.5x ULN or glomerular filtration rate > 50ml/min.
5. ECOG performance status ≤ 3
6. Women of reproductive potential should have a serum pregnancy test or negative urine.
7. Prior signature of the informed consent.

Exclusion Criteria:

1. Voluntary withdrawal from the study.
2. Develop grade 3 or 4 toxicity according to the INH scale.
3. Loss of follow-up

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-10-18 (Estimated); Study Completion 2025-10-18 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 24 months
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first.

SECONDARY OUTCOMES:
complete remission | 24 months
  complete absence of any disease assessed by PET after established treatment
overall survival | 24 months
  status at last follow-up alive or dead

CONTACTS AND LOCATIONS:
Overall Officials: Lauro Amador Medina, Study Director — Hospital regional Alta especialidad Bajío
Locations (1):
- Hospital Regional Alta Especialidad Bajio, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Yes
We have plan to share participant data for metanalysis
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: request by researcher
Access Criteria: request by researcher

REFERENCES:
- [Derived] Barrera Chavez ID, Viloria Alvarez JC, Zendejas Sanchez V, Rodriguez Esquivel A, Alvarez Salinas A, Amador Medina LF. Efficacy of Brentuximab-Vedotin Combined with PD-1 Inhibitors in Relapsed/Refractory Hodgkin Lymphoma with ASCT Consolidation and Maintenance Therapy: A Phase 2 Clinical Trial. Indian J Hematol Blood Transfus. 2026 Jan;42(1):93-99. doi: 10.1007/s12288-025-01986-0. Epub 2025 Feb 17. PMID 41522540